CLINICAL TRIAL: NCT01015677
Title: A Phase IIa, Randomized, Double-Blind, Placebo- and Active-Controlled Study to Examine MK-6913 for the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: A Study of MK-6913 for the Treatment of Hot Flashes in Postmenopausal Women (6913-004)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6913-004; MK-6913-004 (Other: Protocol number)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Moderate to Severe Vasomotor Symptoms in Postmenopausal; Women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-6913 75 mg (Experimental): MK-6913 75 mg capsule and matching placebo for 17β-estradiol 1 mg tablet once daily for 4 weeks (Stage 1 and Stage 2)
  Interventions: Drug: MK-6913; Drug: Placebo to 17-β estradiol
- 17-β estradiol 1 mg (Active Comparator): 17β-estradiol 1 mg tablet and matching placebo for MK-6913 75 mg capsule once daily for 4 weeks (Stage 1 and Stage 2)
  Interventions: Drug: 17-β estradiol; Drug: Placebo to MK-6913
- Placebo (Placebo Comparator): Matching placebo for MK-6913 75 mg capsule and matching placebo for 17β-estradiol 1 mg tablet once daily for 4 weeks (Stage 1 and State 2)
  Interventions: Drug: Placebo to MK-6913; Drug: Placebo to 17-β estradiol
- MK-6913 25 mg (Experimental): MK-6913 25 mg capsule and matching placebo for 17β-estradiol 1 mg tablet once daily for 4 weeks (Stage 2)
  Interventions: Drug: MK-6913 25 mg

INTERVENTIONS:
Drug: MK-6913
  Arms: MK-6913 75 mg
Drug: 17-β estradiol
  Arms: 17-β estradiol 1 mg
Drug: Placebo to MK-6913
  Arms: 17-β estradiol 1 mg; Placebo
Drug: Placebo to 17-β estradiol
  Arms: MK-6913 75 mg; Placebo
Drug: MK-6913 25 mg
  Arms: MK-6913 25 mg

SUMMARY:
This study will assess the safety, tolerability, and efficacy of MK-6913 for the treatment of moderate-to-very-severe vasomotor symptoms (hot flashes or hot flushes) in postmenopausal women. The primary study hypothesis is that one or more doses of MK-6913 will result in a significantly greater reduction from baseline, compared to placebo, in the number of moderate to very severe hot flashes after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Woman with at least 50 moderate to very severe hot flash episodes per week
* Postmenopausal
* Between 45 and 60 years of age if naturally menopausal, or between 35 and 60 if she underwent a bilateral oophorectomy
* Not receiving hormone therapy
* Has had both a normal mammogram and a normal Pap test in the past 6 months
* Generally healthy

Exclusion Criteria:

* A history of cancer, except for certain skin cancers
* Undiagnosed vaginal bleeding or any uterine endometrial disorder
* Currently uses tobacco products, or has used them in the last 6 months
* Has human immunodeficiency virus (HIV)

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2009-12-17 (Actual); Primary Completion 2010-07-30 (Actual); Study Completion 2010-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=6913-004&kw=6913-004&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty sites in the United States, Canada, France, Belgium, New Zealand, and Australia received IRB/ERC approval. Of the 354 participants screened for inclusion, 255 participants were excluded during screening (235 participants did not meet specific exclusion criteria). Ninety-nine participants were randomized for the study.
Pre-assignment Details: The study was terminated at the end of Stage 1 so no participants entered Stage 2 and no participants received MK-6913 25 mg.
Groups:
- MK-6913 75 mg: MK-6913 75 mg and matching placebo for 17β-estradiol 1 mg once daily for 4 weeks
- 17-β Estradiol 1 mg: 17β-estradiol 1 mg and matching placebo for MK-6913 75 mg once daily for 4 weeks
- Placebo: Matching placebo for MK-6913 75 mg and matching placebo for 17β-estradiol 1 mg once daily for 4 weeks
Period: Overall Study
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo
Started | 34 | 32 | 33
Completed | 33 | 28 | 33
Not Completed | 1 | 4 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo | Total
Number analyzed (Participants) | 34 | 32 | 33 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (3.9) | 53.2 (3.9) | 52.2 (4.2) | 52.5 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 33 | 99
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Number of Weekly Moderate to Very Severe Hot Flashes (Excluding Outliers) at Week 4
Description: Hot flashes were recorded in real time and hot flashes recorded retrospectively in the morning and evening reports in a diary day via the Hot Flash e-diary were summed to determine the total number of hot flashes over a diary day. The total number of weekly moderate or worse hot flashes were calculated as the sum of the total number of hot flashes that occur over a diary week (non-missing diary day), divided by the number of days of diary completion, and multiplied by 7 (standardized week). At least 4 non-missing diary days were required to define the total number of weekly moderate or worse hot flashes. Hot flash data was excluded for participants whose number of moderate to severe hot flashes per week were in the top 1% of number of hot flashes reported to exclude any outlier effect.
Time Frame: Baseline and Week 4
Population: The Full Analysis Set (FAS) population consists of all randomized participants who receive at least 1 dose of study treatment, have at least 1 post-randomization observation for the analysis endpoint, and have baseline data for those analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo
Number analyzed (Participants) | 34 | 31 | 33
Percent change | -40.69 [-54.82 to -26.56] | -51.86 [-66.38 to -37.34] | -34.41 [-48.99 to -19.83]
Statistical Analysis 1: Comparison: MK-6913 75 mg vs Placebo; Test type: Superiority or Other; p = 0.488, Longitudinal Data Analysis (LDA); LDA model terms for treatment, week (Weeks 1, 2 and 4), region, and interaction of treatment by week; Differrence in the least squares means = -6.28, 95% CI 2-sided [-24.20 to 11.64]
Statistical Analysis 2: Comparison: 17-β Estradiol 1 mg vs Placebo; Test type: Superiority or Other; p = 0.069, Longitudinal Data Analysis; LDA model with terms for treatment, week (Weeks 1, 2 and 4), region, and interaction of treatment by week; Difference in the least squares means = -17.45, 95% CI 2-sided [-36.28 to 1.38]

2. Primary Outcome: Number of Participants Who Experienced at Least One or More Adverse Events (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 6 weeks
Population: The All-Patients-as Treated (APaT) population is all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo
Number analyzed (Participants) | 34 | 32 | 33
Participants | 17 | 15 | 16

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 4 weeks
Population: The APaT population is all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo
Number analyzed (Participants) | 34 | 32 | 33
Participants | 0 | 1 | 0

4. Secondary Outcome: Percent Change From Baseline in the Weekly Hot Flash Severity Score (Combining Severe and Very Severe Score) at Week 4
Description: Hot flash severity score is calculated by the sum of: the number of mild hot flashes, 2 times number of moderate hot flashes, 3 times the number of severe hot flashes, and 4 times the number of very severe hot flashes. This sum was standardized to a 7-day week if there were any missing days in the e-diary. The severity of each hot flash was recorded by the Hot Flash e-diary.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo
Number analyzed (Participants) | 34 | 31 | 33
Percent change | -39.92 [-54.57 to -25.26] | -45.09 [-60.15 to -30.02] | -33.87 [-48.92 to -18.81]
Statistical Analysis 1: Comparison: MK-6913 75 mg vs Placebo; Test type: Superiority or Other; p = 0.529, Longitudinal Data Analysis (LDA); LDA model includes terms for treatment, week (Weeks 1, 2 and 4), region, and interaction of treatment by week; Differrence in the least squares means = -6.05, 95% CI 2-sided [-25.06 to 12.96]
Statistical Analysis 2: Comparison: 17-β Estradiol 1 mg vs Placebo; Test type: Superiority or Other; p = 0.264, Longitudinal Data Analysis; LDA model includes terms for treatment, week (Weeks 1, 2 and 4), region, and interaction of treatment by week; Difference in the least squares means = -11.22, 95% CI 2-sided [-31.03 to 8.59]

5. Secondary Outcome: Change From Baseline in Follicle-stimulating Hormone (FSH) Level at Week 4
Description: FSH was measured to assess estrogen receptor (ER) selectivity (a biomarker for ERα activity and a pharmacodynamic endpoint).
Time Frame: Baseline and Week 4
Population: The Per-Protocol (PP) population excludes participants due to important deviations from the protocol that may substantially affect the results of the primary and key secondary efficacy endpoints.
Measure: Least Squares Mean (90% Confidence Interval); unit: mIU/mL
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo
Number analyzed (Participants) | 21 | 21 | 28
mIU/mL | -2.02 [-7.91 to 3.87] | -17.48 [-23.08 to -11.89] | -2.96 [-8.54 to 2.62]
Statistical Analysis 1: Comparison: MK-6913 75 mg vs Placebo; Test type: Superiority or Other; p = 0.827, ANCOVA; Analysis of covariance (ANCOVA) with terms for treatment, region, stage of the trial, and baseline value as a covariate in PP population only; Difference in LS means = 0.94, 90% CI 2-sided [-6.19 to 8.07]
Statistical Analysis 2: Comparison: 17-β Estradiol 1 mg vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA with terms for treatment, region, stage of the trial, and baseline value as a covariate in PP population only; Difference in the LS means = -14.52, 90% CI 2-sided [-21.73 to -7.32]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | MK-6913 75 mg | 17-β Estradiol 1 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 17/34 | 15/32 | 16/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-6913 75 mg (N=34) | 17-β Estradiol 1 mg (N=32) | Placebo (N=33)
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Irritability (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Crystal urine (Investigations) | 0 | 0 | 1
Crystal urine present (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0
Protein urine (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 4
Lethargy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 11
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Elevated mood (Psychiatric disorders) | 0 | 1 | 0
Libido increased (Psychiatric disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated at the end of Stage 1 so no participants entered Stage 2 and no participants received MK-6913 25 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.